CLINICAL TRIAL: NCT01414907
Title: VIP (Very Important Patient) Project on Alcohol and Drug Abusers - RCT of Efficacy of the Adding the Health Promotion and Rehabilitation for Treatment of Alcohol and Drug Abusers
Brief Title: Study of Effectiveness of Adding the Health Promotion and Rehabilitation for Treatment for Alcohol and Drug Abusers
Acronym: VIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other); The Swedish Council for Information on Alcohol and Other Drugs (Other); Lund University (Other); Copenhagen University Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Hanne Tønnesen, Professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIP-LU-2011
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Alcoholism; Substance-Related Disorders; Smoking; Chronic Disease; Malnutrition
Keywords: Drinking Behavior; Harm Reduction; Tobacco Use Cessation; Smoking Cessation; Rehabilitation; Health Promotion; Nutrition Therapy; Feeding Behavior; Exercise
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Smoking; Chronic Disease; Malnutrition; Drinking Behavior; Harm Reduction; Tobacco Use Cessation; Smoking Cessation; Feeding Behavior; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Promotion activities (Active Comparator)
  Interventions: Behavioral: Health promotion activities
- No Intervention (No Intervention)

INTERVENTIONS:
Behavioral: Health promotion activities — Counselled activities on tobacco smoking secession, diet correlation and physical activities
  Other Names: smoking secession; physical activity; diet
  Arms: Health Promotion activities

SUMMARY:
The purpose of this study is to evaluate the effect of adding the Health Promotion activities and rehabilitation to the usual alcohol and drug interventions on the outcome for alcohol and drug abusers compared to the usual intervention alone.

DETAILED DESCRIPTION:
Background: Alcohol and drug abuse are followed by tremendous physical, psychological and social problems as well as early death. Heavy smoking, poor nutrition, physical inactivity and chronic diseases (co-morbidity) are often part of these problems and illnesses.

There seems to be a large potential for a better outcome by including smoking cessation, physical training, diet and nutrition as well as co-morbidity in a multi-disciplinary setting - a potential not used yet. This Very Integrated Program (VIP) is inspired from the rehabilitation offered to patients with chronic diseases and surgical patients having a likewise unhealthy lifestyle and similar co-morbidity.

Aim: to evaluate the effect of adding the VIP program to the usual alcohol and drug intervention on the outcome for alcohol and drug abusers compared to the usual intervention alone.

The VIP project consists of 3 steps:

1. To map the health status and estimate the potential improvement for 400 alcohol and drug abusers
2. To pilot test the VIP program
3. To evaluate it compared to the daily routines for 260 alcohol and drug abusers with a poor health status in a randomised controlled trial.

Main outcome: Change from abuser to non-abuser. Secondary outcomes are health status; quality of life, use of health services, time return to work (or similar activity level), harm reduction, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* alcohol or drug dependency

Exclusion Criteria:

* withdrawal of informed consent
* missing competence to give informed consent
* pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from abuser to non-abuser | 6 weeks, 3, 6, 9, 12 and 24 months

SECONDARY OUTCOMES:
Health status | 6 weeks, 3, 6, 9, 12 and 24 months
Quality of life | 6 weeks, 3,6,9,12 and 24 months
Harm reduction | 6 weeks, 3,6,9,12 and 24 months
Cost-effectiveness | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Tønnesen, MD, PhD, Principal Investigator — WHO-CC, Bispebjerg University Hopital, Copenhagen, Denmark
Locations (1):
- Addiction Center Malmo, Psychiatry Skane, Skane University Hospital, Malmo, Skåne County, Sweden

REFERENCES:
- [Background] Tønnesen H, Hovhannisyan K, Ehrnström M, Skibelund D, Kovacs J, Thornqvist K, Skagert E. Co-morbidity in drug and alcohol addicts - a VIP project. 19th International Conference on Health Promotion Hospitals and Health Services, June 2011, Turku, Finland
- See also: VIP project — http://www.med.lu.se/hvs/alkoholforskning/medarbetare/hanne_toennesen/vip_projektet